CLINICAL TRIAL: NCT07281664
Title: Transarterial Chemoembolization Combined With Low-Dose Bevacizumab Plus Atezolizumab as First-Line Treatment for Unresectable Hepatocellular Carcinoma: A Phase II, Single-Arm Clinical Trial
Brief Title: Transarterial Chemoembolization With Low-Dose Bevacizumab Plus Atezolizumab as First-Line Treatment for Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Huang Mingsheng, The director of Department of Interventional Radiology, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: II2025-380-01
Record Dates: First submitted 2025-11-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Transarterial Chemoembolization
Keywords: Hepatocellular Carcinoma; Transarterial chemoembolization; Bevacizumab; Atezolizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE + LDBev + Atezo (Experimental): Participants in this single-arm study will receive a combination treatment consisting of transarterial chemoembolization (TACE) followed by systemic therapy with low-dose bevacizumab and atezolizumab. TACE will be performed as the locoregional therapy to control intrahepatic tumors, after which bevacizumab and atezolizumab will be administered to inhibit angiogenesis and enhance antitumor immune activity. All participants will be treated according to the study protocol to evaluate the safety and clinical activity of this integrated therapeutic approach for unresectable hepatocellular carcinoma.
  Interventions: Procedure: Transarterial chemoembolization (TACE); Drug: bevacizumab and atezolizumab

INTERVENTIONS:
Procedure: Transarterial chemoembolization (TACE) — The intervention consisted of TACE combined with low-dose bevacizumab and atezolizumab. TACE was performed within 30 days before or after systemic therapy. The choice between conventional TACE and DEB-TACE was determined by interventional radiologists, as both techniques show comparable efficacy. For DEB-TACE, epirubicin-loaded microspheres were used; for conventional TACE, an epirubicin-lipiodol emulsion was prepared. In all cases, the tumor-feeding artery was super-selectively catheterized, and embolization was performed to complete arterial stasis using gelatin sponge particles.
  Following TACE-induced ischemic and cytotoxic tumor control, patients received systemic therapy consisting of low-dose bevacizumab to attenuate post-TACE angiogenic rebound and atezolizumab to enhance antitumor immune activation. This sequential combination of locoregional therapy and dual-agent systemic therapy constitutes a distinct intervention compared with standard TACE or systemic therapy alone.
Drug: bevacizumab and atezolizumab — Low dose bevacizumab and atezolizumab

SUMMARY:
This study aims to evaluate the safety and effectiveness of a combined treatment for patients with unresectable hepatocellular carcinoma (HCC), a type of liver cancer that cannot be removed by surgery. The treatment includes transarterial chemoembolization (TACE), which delivers chemotherapy directly into the liver tumor, together with low-dose bevacizumab and atezolizumab, two medicines that help the immune system fight cancer and inhibit tumor blood vessel growth.

All participants in this study will receive the same combination treatment as their first-line therapy. The study will observe how well the tumor responds, how long the treatment can control the cancer, and what side effects may occur. The goal is to learn whether this combined approach can provide clinical benefit and improve outcomes for patients with advanced, unresectable liver cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is often diagnosed at an advanced stage, when surgical treatment is no longer possible. Transarterial chemoembolization (TACE) is widely used for locoregional control, but many patients eventually experience tumor progression due to treatment-related hypoxia and activation of pro-angiogenic pathways. Combining TACE with systemic therapies that block angiogenesis and enhance antitumor immunity may help overcome these limitations.

Bevacizumab, an anti-VEGF antibody, reduces tumor angiogenesis and may counteract the surge in VEGF that occurs after TACE. Atezolizumab, an immune checkpoint inhibitor, strengthens the immune response against cancer cells. Using low-dose bevacizumab together with atezolizumab may help maximize immunotherapy benefit while minimizing toxicity, especially when administered after TACE.

This single-arm Phase II study is designed to investigate whether integrating TACE with low-dose bevacizumab and atezolizumab as first-line treatment can improve clinical outcomes in patients with unresectable HCC. The study will evaluate tumor control, treatment duration, and safety in real-world clinical settings. The findings may provide evidence to support a multimodal treatment strategy that targets both the tumor vasculature and the immune microenvironment, potentially offering a more effective option for patients with advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between18 and 75 years;
* Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
* Child-Pugh class A;
* Eastern Cooperative Group performance status (ECOG) score of 0-1;
* No prior systemic therapy for HCC.
* Adequate hematologic and end-organ function;
* At least one measurable intrahepatic target lesion.

Exclusion Criteria:

* Diffuse HCC;
* Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes (confirmed by histology, or pathology) are not eligible;
* Evidence of extrahepatic spread (EHS);
* Any condition representing a contraindication to TACE or I-125 seeds brachytherapy as determined by the investigators;
* Evidence or history of bleeding diathesis or any hemorrhage or bleeding event >CTCAE grade 3 within 4 weeks prior to randomization;
* Active or history of autoimmune disease or immune deficiency;
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding;
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment;
* Evidence of bleeding diathesis or significant coagulopathy;
* Pregnant or breastfeeding females;
* Significant cardiovascular disease;
* Severe infection, such as active tuberculosis;
* Serious medical comorbidities;
* History of organ or cells transplantation;
* History of other uncurable malignancies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Time from randomization to disease progression (mRECIST) or death from any cause, whichever occurred first.

OTHER OUTCOMES:
Objective response rate (ORR) | 2 years
  The percentage of patients who had a best overall tumor response rating of CR and PR (mRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Mingsheng Huang, M.D. & Ph.D, Principal Investigator — Department of Interventional Radiology, The Third Affiliated Hospital of Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may be shared upon reasonable request. Any data sharing will be discussed and agreed upon with the corresponding author to ensure that it complies with ethical, regulatory, and institutional requirements.